CLINICAL TRIAL: NCT06956729
Title: Guided Growth in Spastic Hip - Multicenter Study (GGSH-MC)
Brief Title: Multicenter Trial of Proximal Femoral Guided Growth in Children With CP and Hips at Risk of Dislocation (GGSH-MC)
Acronym: GGSH-MC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación para la investigación biomética Hospital Infantil Universitario Niño Jesús (Other)
Collaborators: Hospital Sant Joan de Deu (Other); Salamanca University Hospital (Other); Complexo Hospitalario Universitario de A Coruña (Other); Hospital General Universitario Gregorio Marañon (Other); Hospital Universitario de Canarias (Other); Hospital Universitario Central de Asturias (Other); Hospital Son Espases (Other); Hospital Universitario 12 de Octubre (Other); Hospital Vall d'Hebron (Other); Hospital Universitario Virgen Macarena (Other); Hospital Miguel Servet (Other); Hospital Donostia (Other); Hospitales Universitarios Virgen del Rocío (Other); Complejo Hospitalario de Navarra (Other); Hospital Universitario Ramon y Cajal (Other); Hospital Universitario Torrecárdenas (Other)
Responsible Party: Principal Investigator, María Galán Olleros, Specialist in Orthopedic Surgery and Traumatology., Hospital Infantil Universitario Niño Jesús, Madrid, Spain
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.I.R-0041-24; PR-PI24-00016 (Other Grant/Funding Number: European Paediatric Orthopaedic Society (EPOS))
Record Dates: First submitted 2025-03-19; First posted 2025-05-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Cerebral Palsy
Keywords: Proximal Femoral Guided Growth; Randomized Controlled Trial; Spastic Hip; Hip Dislocation
MeSH Terms: conditions — Cerebral Palsy; Hip Dislocation

STUDY DESIGN:
Intervention Model Description: This study is a prospective, multicenter, randomized controlled trial (RCT) with two parallel groups, using cluster randomization to minimize inter-center variability in surgical techniques and postoperative care. Centers are assigned to either the experimental group (PFGG + standard prophylactic treatment) or the control group (standard prophylactic treatment alone). Conducted across specialized pediatric orthopedic centers, the study includes a one-year enrollment period, followed by a 24-month structured follow-up with standardized clinical and radiographic assessments at 3 weeks, 6 weeks, 6, 12, 18, and 24 months. The intervention is single-blinded, ensuring radiographic assessors and outcome evaluators remain unaware of group allocation to reduce bias. Data will be analyzed using intention-to-treat principles to account for any deviations from the assigned interventions.
Masking Description: Functional outcome evaluators and data analysts will be blinded to group allocation. Although radiographic assessors cannot be fully blinded due to visible hardware, they will be independent and follow standardized protocols to ensure objectivity. Treating surgeons and caregivers will not be blinded due to the nature of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PFGG + Standard Treatment (Experimental Group A) (Experimental): Participants in this arm will receive Proximal Femoral Guided Growth (PFGG) in addition to standard prophylactic treatment for hips at risk of dislocation (HRD).
  The standard treatment may include adductor tenotomy (percutaneous or open) and psoas tenotomy (intrapelvic or at the lesser trochanter) as indicated.
  Surgery will be performed under general anesthesia, and postoperative immobilization will follow institutional protocols, including the use of a hip abduction wedge, knee immobilizers, and ankle-foot orthoses (AFO) as required.
  Follow-up will include standardized clinical, functional, and radiographic assessments at 3 weeks, 6 weeks, 6 months, 12 months, 18 months, and 24 months postoperatively.
  Interventions: Procedure: Proximal Femoral Guided Growth.; Procedure: Standard prophylactic treatment for Hips at Risk of Dislocation.
- Standard Treatment Only (Control Group B) (Active Comparator): Participants in this arm will receive standard prophylactic treatment for HRD without PFGG.
  This may include adductor and/or psoas tenotomies based on clinical indication, performed under general anesthesia.
  Postoperative care will be identical to the experimental group, with standard immobilization using a hip abduction wedge, knee immobilizers, and AFOs as needed.
  The follow-up schedule and outcome assessments will be identical to the experimental group, ensuring consistency in data collection.
  Interventions: Procedure: Standard prophylactic treatment for Hips at Risk of Dislocation.

INTERVENTIONS:
Procedure: Proximal Femoral Guided Growth. — Proximal Femoral Guided Growth (PFGG) is performed under general anesthesia with the patient in a supine position on a radiolucent table. The surgical field is prepared from the abdomen to the feet. Anatomical landmarks on the femur and femoral neck are marked to guide the procedure.
  A smooth guidewire (4.0-7.0 mm) is introduced parallel to the table and advanced to the lateral quarter of the femoral neck.
  A 1-2 cm incision is made along the lateral femur, allowing access to the vastus lateralis muscle.
  Fluoroscopic control is used to ensure precise guidewire placement in the proximal femoral epiphysis in both anteroposterior (AP) and lateral views.
  The lateral cortex is drilled, and a fully threaded cannulated screw is inserted, ensuring at least three threads reach the epiphysis for effective growth modulation.
  Final fluoroscopic verification is performed to confirm proper screw placement and rule out joint penetration. Continuous fluoroscopy is used if necessary.
  The guidewire is r
  Other Names: Guided Growth Surgery; Proximal Femoral Epiphysiodesis; Proximal Femoral Hemiepiphysiodesis
  Arms: PFGG + Standard Treatment (Experimental Group A)
Procedure: Standard prophylactic treatment for Hips at Risk of Dislocation. — Both groups will receive standard prophylactic treatment for HRD, which consists of soft tissue release procedures based on clinical indication and functional level (GMFCS classification):
  Adductor Tenotomy - Percutaneous or open technique, depending on contracture severity.
  Psoas Tenotomy - Intrapelvic approach for GMFCS levels I-III and IV (ambulatory). Lesser trochanter approach for GMFCS levels IV-V (non-ambulatory). Additional tenotomies may be performed as needed, targeting muscles contributing to hip displacement and contractures.
  Botulinum toxin type A may be administered to specific muscle groups if clinically indicated.
  Postoperative immobilization includes:
  Hip abduction wedge Knee immobilizers in extension Ankle-foot orthoses (AFOs), based on individual patient needs
  The goal of this intervention is to reduce spastic muscle imbalance, improve hip stability, and delay or prevent hip dislocation in children with spastic CP and HRD.

SUMMARY:
The Guided Growth in Spastic Hip Multicenter Study (GGSH-MC) is a prospective, multicenter, randomized controlled trial that aims to evaluate the mid-term outcomes of Proximal Femoral Guided Growth (PFGG) in children with spastic cerebral palsy (CP) and hips at risk of dislocation (HRD). Hip dislocation is a common and severe complication in children with CP, especially those who are non-ambulatory, with a reported risk of 70-90%.

The trial includes children aged 3 to 8 years with spastic CP and HRD, defined by a migration percentage (MP) between 30% and 60%. Participants will be cluster-randomized by center into two parallel groups:

* Experimental Group: Standard prophylactic treatment for HRD + PFGG
* Control Group: Standard prophylactic treatment for HRD only

PFGG involves insertion of a fully threaded cannulated screw across the lateral cortex and proximal femoral epiphysis under fluoroscopic guidance, with the aim of modulating growth to improve hip containment. All patients will also receive standard soft tissue surgery (adductor and/or psoas tenotomies), as clinically indicated.

Follow-up will include clinical, radiographic, and functional assessments at 3 and 6 weeks, and at 6, 12, 18, and 24 months post-intervention. The study will include a 1-year inclusion period and a 2-year follow-up, concluding in October 2027.

Primary outcome measures include radiographic indicators of hip displacement. Secondary outcomes include functional scores, complication rates, and need for further surgery. A total of 42 participants (21 per group) will provide 80% power to detect significant differences at a 0.05 significance level. Analyses will be performed using intention-to-treat principles, with subgroup and multivariate analyses to explore modifying factors.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is the leading cause of severe physical disability in childhood, with a prevalence of 1.6 per 1,000 live births in developed countries. Spastic CP, affecting 75% of patients, often leads to progressive musculoskeletal deformities due to muscle imbalance, particularly around the hip joint. Hip dysplasia is the second most common deformity, and if untreated, can progress to dislocation, especially in non-ambulatory children (GMFCS IV-V), where risk exceeds 70%.

Hip displacement in CP is attributed to spasticity of the adductors and flexors, growth-related deformities such as coxa valga and acetabular dysplasia, and limited weight-bearing. These changes can impair function, sitting tolerance, hygiene, and quality of life. Current strategies emphasize surveillance and early intervention for hips at risk of dislocation (HRD), including soft tissue surgery. However, recurrence remains high, and reconstructive surgery, while effective, is invasive and associated with significant morbidity.

Proximal Femoral Guided Growth (PFGG) is a minimally invasive technique involving medial hemiepiphysiodesis with a cannulated screw to modulate proximal femoral growth and improve containment. Though early outcomes are promising, prospective multicenter evidence is limited.

This study is a prospective, multicenter, randomized controlled trial using cluster randomization by center to compare PFGG + standard treatment versus standard treatment alone. Children aged 3-8 years with spastic CP and HRD (MP 30-60%) will be included. The primary outcome is radiographic containment. Secondary outcomes include functional scores, pain, complications, and reintervention rates. Follow-up spans 24 months.

All surgeries follow a standardized protocol. Postoperative care includes early mobilization, use of hip abduction wedge, and physical therapy. Sample size is calculated for 80% power to detect a difference in dislocation rates, requiring 42 subjects. Data will be collected using standardized CRFs and managed centrally under SEOP oversight. Adverse events will be systematically recorded.

The study has IRB approval and complies with ISO 14155, GDPR, and the Helsinki Declaration. Funding is provided by the 2023 EPOS Research Grant (€10,000). Results will be published regardless of outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 3 to 8 years.
* Diagnosis of predominantly spastic cerebral palsy (CP).
* Any functional level according to the GMFCS.
* Hips at risk of dislocation (HRD), unilateral or bilateral, defined by a migration percentage (MP) between 30% and 60%.

Exclusion Criteria:

* Children with predominantly hypotonic or dystonic types of CP.
* Children with neuromuscular conditions other than CP.
* Children with high surgical/anesthetic risk.
* Documented history of reconstructive or palliative hip surgery.

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Migration percentage (MP). Radiological | Pre-surgery; 3 weeks; 6, 12, 18, and 24 months post-surgery
  Percentage of the femoral head lateral to Perkins line on standardized AP pelvic radiograph. Unit of Measure: Percentage (%)
Pelvic Obliquity (PO). Radiological | Pre-surgery; 3 weeks; 6, 12, 18, and 24 months post-surgery.
  Angle between the horizontal line and the line joining both iliac crests on AP pelvic radiograph. Unit of Measure: Degrees (°)
Migration Percentage Adjusted for Pelvic Obliquity (PAMP). Radiological | Pre-surgery; 3 weeks; 6, 12, 18, and 24 months post-surgery.
  Modified MP accounting for pelvic tilt, measured on AP pelvic radiograph. Unit of Measure: Percentage (%)
Acetabular Index (AI). Radiological | Pre-surgery; 3 weeks; 6, 12, 18, and 24 months post-surgery.
  Angle formed between Hilgenreiner's line and a line along the acetabular roof. Unit of Measure: Degrees (°)
Center-Edge Angle (CEA). Radiological | Pre-surgery; 3 weeks; 6, 12, 18, and 24 months post-surgery.
  Angle between vertical line through femoral head center and a line to lateral acetabular edge. Unit of Measure: Degrees (°)
Hilgenreiner Epiphyseal Angle (HEA). Radiological | Pre-surgery; 3 weeks; 6, 12, 18, and 24 months post-surgery.
  Angle between Hilgenreiner's line and a line along the proximal femoral physis. Unit of Measure: Degrees (°)

SECONDARY OUTCOMES:
Patient characteristics. Age | At time of surgery
  Chronological age of the patient at the time of surgery. Unit of measure: years
Patient characteristics. Sex | Pre-surgery
  Biological sex of participant. Unit of Measure: Male/Female
Patient characteristics. Gross Motor Function Classification System level (GMFCS) | Pre-surgery
  GMFCS level will be recorded to classify gross motor function. The GMFCS has five levels (I to V), with higher levels indicating more severe motor impairment.
  Unit of measure: scale (I to V)
Patient characteristics. Weight | Pre-surgery
  Weight of the patient measured using a calibrated scale during the pre-surgical evaluation.
  Unit of measure: kilograms (kg)
Patient characteristics. Orthopedic comorbidities | Pre-surgery
  Presence or absence of orthopedic comorbidities such as scoliosis and knee flexion contractures will be assessed.
Patient characteristics. Respiratory disorders or gastrointestinal issues | Pre-surgery
  Presence or absence of relevant medical comorbidities, including epilepsy, respiratory disorders (e.g., obstructive sleep apnea, tracheostomy), and gastrointestinal disorders (e.g., gastrostomy), will be recorded.
Patient characteristics. Medication use | Pre-surgery
  Current use of any medication will be recorded as a categorical variable (yes/no), along with medication type if applicable.
Clinical variables. Pain | Immediately after surgery; 3 and 6 weeks; 6, 12, 18, and 24 months post-surgery
  Pain will be assessed using the Visual Analog Scale (VAS), a 10-cm horizontal line ranging from "no pain" to "worst imaginable pain." Higher scores indicate greater pain intensity.
  Unit of measure: scale (0-10)
Clinical variables. Analgesic needs | Immediately after surgery; 3 and 6 weeks; 6, 12, 18, and 24 months post-surgery
  Analgesic requirements will be recorded based on caregiver reports.
  Categorical: first-line analgesics (e.g., Ibuprofen, Paracetamol [Acetaminophen], Metamizole), second-line analgesics (e.g., mild opioids like Tramadol), or third-line analgesics (e.g., strong opioids such as morphine and fentanyl).
Clinical variables. Hip abduction in flexion | Pre-surgery; at 6 weeks, 6 months, 12, 18, and 24 months
  Hip abduction in flexion will be measured in degrees during standardized physical examination. Unit of Measure: Degrees (º)
Clinical variables. Hip abduction in extension | Pre-surgery; at 6 weeks, 6 months, 12, 18, and 24 months
  Hip abduction in extension will be measured in degrees during standardized physical examination. Unit of Measure: Degrees (º)
Clinical variables. Hip flexion contracture >20° | Pre-surgery; at 6 weeks, 6 months, 12, 18, and 24 months
  Presence or absence of hip flexion contracture greater than 20 degrees will be recorded during physical examination. Yes/no
Clinical variables. Galeazzi sign | Pre-surgery; at 6 weeks, 6 months, 12, 18, and 24 months
  The Galeazzi sign will be assessed to detect femoral shortening as a clinical indicator of limb length discrepancy. Presence or absence will be recorded.
Clinical variables. Pelvic obliquity | Pre-surgery; at 6 weeks, 6 months, 12, 18, and 24 months
  Pelvic obliquity will be assessed clinically during physical examination and recorded as present or absent.
Functional variables | Pre-surgery; 12 and 24 months
  The Caregiver Priorities and Child Health Index of Life with Disabilities (CPCHILD) questionnaire will be completed. It is a validated measure of health-related quality of life for children with severe disabilities. Units on a scale (0-100; higher = better)
Concomitant treatment. Physiotherapy Frequency Per Week | At 6 weeks; 6, 12, 18, and 24 months
  Frequency of physiotherapy: Number of Physiotherapy Sessions per Week. Sessions per week.
Concomitant treatment. Orthoses Use | At 6 weeks; 6, 12, 18, and 24 months
  Use of orthoses: Number of hours per day the participant uses orthotic devices (e.g., hip abduction orthoses, scoliosis braces. Unit of Measure: Hours per day.
Concomitant treatment. Weight-Bearing Activity Time | At 6 weeks; 6, 12, 18, and 24 months
  Time Spent in Weight-Bearing Activities per Day. Unit of Measure: Minutes per day.
Concomitant treatment. Participation in Complementary Therapies | At 6 weeks; 6, 12, 18, and 24 months
  Participation in Complementary Therapies such as Hydrotherapy, hippotherapy, or other specified therapies. Unit of Measure: Yes/No.
Safety variables and parameters. Clinical complications | Immediately after surgery; 3 weeks; 6 weeks; 6 months; 12 months; 18 months; 24 months post-surgery
  Wound dehiscence, hematoma, superficial or deep infection. New symptoms not present before surgery will also be evaluated, such as pain, hip mobility limitations or stiffness, insomnia, constipation, irritability, etc.
  Unit of Measure of all the above: Participants
Safety variables and parameters. Radiological complications | Immediately after surgery; 3 weeks; 6 weeks; 6 months; 12 months; 18 months; 24 months post-surgery
  Loosening of epiphyseal screws, peri-implant fracture, implant breakage, progression of hip displacement, avascular necrosis of the femoral head, chondrolysis, etc.
  Unit of Measure: Number of participants
Safety variables and parameters. Functional complications | Immediately after surgery; 3 weeks; 6 weeks; 6 months; 12 months; 18 months; 24 months post-surgery
  Intolerance to sitting, supine or lateral positioning, difficulty in perineal care, hygiene, or dressing.
  Unit of Measure of all the above: Participants
Safety variables and parameters. Clavien-Dindo-Sink surgical complications classification | Immediately after surgery; 3 weeks; 6 weeks; 6 months; 12 months; 18 months; 24 months post-surgery
  Complications will be classified according to the modified Clavien-Dindo-Sink surgical complications classification. Unit of Measure: Grade (Ordinal)
Other variables. Surgical time | Perioperative (intraoperative)
  Measured from skin incision to closure, quantified in minutes
Other variables. Postoperative hospital stay | From surgery to discharge
  Measured in days, with the day of surgery as day 0.
Other variables. Time to comfortable wheelchair sitting | At 3 weeks post-surgery
  Number of days until the patient can sit comfortably in a wheelchair after surgery (day 0), as reported by primary caregivers.
Other variables. Time until pain-free perineal care and hygiene | Assessed at 3 weeks post-surgery
  Number of days until the patient can perform perineal care and hygiene without pain post-surgery (day 0), reported by primary caregivers during follow-up.
Other variables. Time to initiation of pain-free physiotherapy | Assessed at 3 weeks post-surgery
  Number of days from the surgical intervention (day 0) until the patient can begin physiotherapy without pain, as reported by primary caregivers during follow-up visits.

CONTACTS AND LOCATIONS:
Overall Officials: María Galán Olleros, MD, Principal Investigator — Hospital Infantil Universitario Niño Jesús, Madrid
Locations (16):
- Spain (16):
  - H. Materno Inf. Teresa Herrera, A Coruña, A Coruña
  - Hospital Universitario Torrecárdenas Almeria, Almería, Andalusia
  - H.U. Virgen Macarena Sevilla, Seville, Andalusia
  - H.U. Virgen Del Rocio, Seville, Andalusia
  - Ihp-Orthopediatica Sevilla, Seville, Andalusia
  - H. Universitari Son Espases, Palma, Balearic Islands
  - H. Universitario de Salamanca, Salamanca, Castille and León
  - H. Sant Joan de Deu, Barcelona, Catalonia
  - Donostia University Hospital, Donostia / San Sebastian, Gipuzkoa
  - H. U. Gregorio Marañón, Madrid, Madrid
  - Hospital Infantil Universitario Niño Jesús, Madrid, Madrid
  - Hospital Universitario Ramón Y Cajal, Madrid, Madrid
  - Hospital Universitario Doce de Octubre, Madrid, Madrid
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - H.U. Central de Asturias, Oviedo, Principality of Asturias
  - H. Univ. de Canarias, Santa Cruz de Tenerife, Santa Cruz de Tenerife

IPD SHARING:
Plan to Share IPD: Yes
Participant data will be processed in accordance with current data protection legislation, including Organic Law 3/2018, of December 5, on Data Protection and Digital Rights, and the European Regulation (EU) 2016/679 (GDPR). This means that:
  * The data controller is the Sponsor: SEOP Neuro-Orthopedics Working Group (Spanish Society of Pediatric Orthopedics). Data will be shared among study centers for statistical purposes only.
  * Personal information is stored in medical records.
  * Data will not leave the EU and will remain confidential.
  * Patients may exercise their data rights and file complaints.
  * Patients' names will not appear in any publications.
Supporting Information: Study Protocol, SAP
Time Frame: Individual participant data and supporting documentation (Study Protocol and Statistical Analysis Plan) will be available beginning 6 months after the publication of the primary results and will remain accessible for 5 years. Data access will be limited to approved researchers under controlled conditions for statistical purposes only.
Access Criteria: * The data controller is the Sponsor: SEOP Group (Sociedad Española de Ortopedia Pediátrica). Data will be shared among study centers for statistical purposes only.
  * Each participant: personal information will be stored in their medical record. Only the principal investigator and collaborators will be able to identify participants, as they will manage the database linking the assigned codes to each individual. Only health authorities or the Ethics Committee will have access to this information, ensuring confidentiality.

REFERENCES:
- [Background] Kiapekos N, Brostrom E, Hagglund G, Astrand P. Primary surgery to prevent hip dislocation in children with cerebral palsy in Sweden: a minimum 5-year follow-up by the national surveillance program (CPUP). Acta Orthop. 2019 Oct;90(5):495-500. doi: 10.1080/17453674.2019.1627116. Epub 2019 Jun 18. PMID 31210072
- [Background] Shore BJ, Yu X, Desai S, Selber P, Wolfe R, Graham HK. Adductor surgery to prevent hip displacement in children with cerebral palsy: the predictive role of the Gross Motor Function Classification System. J Bone Joint Surg Am. 2012 Feb 15;94(4):326-34. doi: 10.2106/JBJS.J.02003. PMID 22336971
- [Background] Hwang M, Kuroda MM, Tann B, Gaebler-Spira DJ. Measuring care and comfort in children with cerebral palsy: the care and comfort caregiver questionnaire. PM R. 2011 Oct;3(10):912-9. doi: 10.1016/j.pmrj.2011.05.017. PMID 21852220
- [Background] Hagglund G, Goldring M, Hermanson M, Rodby-Bousquet E. Pelvic obliquity and measurement of hip displacement in children with cerebral palsy. Acta Orthop. 2018 Dec;89(6):652-655. doi: 10.1080/17453674.2018.1519104. Epub 2018 Oct 17. PMID 30326758
- [Background] Narayanan UG, Fehlings D, Weir S, Knights S, Kiran S, Campbell K. Initial development and validation of the Caregiver Priorities and Child Health Index of Life with Disabilities (CPCHILD). Dev Med Child Neurol. 2006 Oct;48(10):804-12. doi: 10.1017/S0012162206001745. PMID 16978459
- [Background] Birkenmaier C, Jorysz G, Jansson V, Heimkes B. Normal development of the hip: a geometrical analysis based on planimetric radiography. J Pediatr Orthop B. 2010 Jan;19(1):1-8. doi: 10.1097/BPB.0b013e32832f5aeb. PMID 19829156
- [Background] Foroohar A, McCarthy JJ, Yucha D, Clarke S, Brey J. Head-shaft angle measurement in children with cerebral palsy. J Pediatr Orthop. 2009 Apr-May;29(3):248-50. doi: 10.1097/BPO.0b013e31819bceee. PMID 19305274
- [Background] Southwick WO. Osteotomy through the lesser trochanter for slipped capital femoral epiphysis. J Bone Joint Surg Am. 1967 Jul;49(5):807-35. No abstract available. PMID 6029256
- [Background] Tonnis D. Normal values of the hip joint for the evaluation of X-rays in children and adults. Clin Orthop Relat Res. 1976 Sep;(119):39-47. PMID 954321
- [Background] Reimers J. The stability of the hip in children. A radiological study of the results of muscle surgery in cerebral palsy. Acta Orthop Scand Suppl. 1980;184:1-100. doi: 10.3109/ort.1980.51.suppl-184.01. No abstract available. PMID 6930145
- [Background] Onimus M, Allamel G, Manzone P, Laurain JM. Prevention of hip dislocation in cerebral palsy by early psoas and adductors tenotomies. J Pediatr Orthop. 1991 Jul-Aug;11(4):432-5. doi: 10.1097/01241398-199107000-00002. PMID 1860938
- [Background] Lebe M, van Stralen RA, Buddhdev P. Guided Growth of the Proximal Femur for the Management of the 'Hip at Risk' in Children with Cerebral Palsy-A Systematic Review. Children (Basel). 2022 Apr 25;9(5):609. doi: 10.3390/children9050609. PMID 35626786
- [Background] Hsu PJ, Wu KW, Lee CC, Lin SC, Kuo KN, Wang TM. Does screw position matter for guided growth in cerebral palsy hips? Bone Joint J. 2020 Sep;102-B(9):1242-1247. doi: 10.1302/0301-620X.102B9.BJJ-2020-0340.R1. PMID 32862682
- [Background] Portinaro N, Turati M, Cometto M, Bigoni M, Davids JR, Panou A. Guided Growth of the Proximal Femur for the Management of Hip Dysplasia in Children With Cerebral Palsy. J Pediatr Orthop. 2019 Sep;39(8):e622-e628. doi: 10.1097/BPO.0000000000001069. PMID 31393306
- [Background] Hsieh HC, Wang TM, Kuo KN, Huang SC, Wu KW. Guided Growth Improves Coxa Valga and Hip Subluxation in Children with Cerebral Palsy. Clin Orthop Relat Res. 2019 Nov;477(11):2568-2576. doi: 10.1097/CORR.0000000000000903. PMID 31425278
- [Background] Lee WC, Kao HK, Yang WE, Ho PC, Chang CH. Guided Growth of the Proximal Femur for Hip Displacement in Children With Cerebral Palsy. J Pediatr Orthop. 2016 Jul-Aug;36(5):511-5. doi: 10.1097/BPO.0000000000000480. PMID 25887815
- [Background] Chou PC, Huang YC, Hsueh CJ, Lin JG, Chu HY. Retrospective study using MRI to measure depths of acupuncture points in neck and shoulder region. BMJ Open. 2015 Jul 29;5(7):e007819. doi: 10.1136/bmjopen-2015-007819. PMID 26224017
- [Background] Shaw KA, Hire JM, Cearley DM. Salvage Treatment Options for Painful Hip Dislocations in Nonambulatory Cerebral Palsy Patients. J Am Acad Orthop Surg. 2020 May 1;28(9):363-375. doi: 10.5435/JAAOS-D-19-00349. PMID 31663909
- [Background] Shore BJ, Graham HK. Management of Moderate to Severe Hip Displacement in Nonambulatory Children with Cerebral Palsy. JBJS Rev. 2017 Dec;5(12):e4. doi: 10.2106/JBJS.RVW.17.00027. No abstract available. PMID 29256976
- [Background] Shrader MW, Wimberly L, Thompson R. Hip Surveillance in Children With Cerebral Palsy. J Am Acad Orthop Surg. 2019 Oct 15;27(20):760-768. doi: 10.5435/JAAOS-D-18-00184. PMID 30998565
- [Background] Hagglund G, Andersson S, Duppe H, Lauge-Pedersen H, Nordmark E, Westbom L. Prevention of dislocation of the hip in children with cerebral palsy. The first ten years of a population-based prevention programme. J Bone Joint Surg Br. 2005 Jan;87(1):95-101. PMID 15686244
- [Background] Ramstad K, Jahnsen RB, Terjesen T. Severe hip displacement reduces health-related quality of life in children with cerebral palsy. Acta Orthop. 2017 Apr;88(2):205-210. doi: 10.1080/17453674.2016.1262685. Epub 2016 Nov 28. PMID 27892753
- [Background] Wawrzuta J, Willoughby KL, Molesworth C, Ang SG, Shore BJ, Thomason P, Graham HK. Hip health at skeletal maturity: a population-based study of young adults with cerebral palsy. Dev Med Child Neurol. 2016 Dec;58(12):1273-1280. doi: 10.1111/dmcn.13171. Epub 2016 Jun 17. PMID 27312016
- [Background] Jung NH, Pereira B, Nehring I, Brix O, Bernius P, Schroeder SA, Kluger GJ, Koehler T, Beyerlein A, Weir S, von Kries R, Narayanan UG, Berweck S, Mall V. Does hip displacement influence health-related quality of life in children with cerebral palsy? Dev Neurorehabil. 2014 Dec;17(6):420-5. doi: 10.3109/17518423.2014.941116. Epub 2014 Jul 24. PMID 25057804
- [Background] Cornell MS. The hip in cerebral palsy. Dev Med Child Neurol. 1995 Jan;37(1):3-18. doi: 10.1111/j.1469-8749.1995.tb11928.x. No abstract available. PMID 7828785
- [Background] Bagg MR, Farber J, Miller F. Long-term follow-up of hip subluxation in cerebral palsy patients. J Pediatr Orthop. 1993 Jan-Feb;13(1):32-6. doi: 10.1097/01241398-199301000-00007. PMID 8416350
- [Background] Kerr Graham H, Selber P. Musculoskeletal aspects of cerebral palsy. J Bone Joint Surg Br. 2003 Mar;85(2):157-66. doi: 10.1302/0301-620x.85b2.14066. No abstract available. PMID 12678344